CLINICAL TRIAL: NCT07179679
Title: A Phase I Clinical Study to Evaluate the Safety and Pharmacokinetics of TQB2934 Subcutaneous Preparation for Injection in Subjects With Malignant Plasma Cell Tumors
Brief Title: A Clinical Study Assessing the Subcutaneous Formulation of TQB2934 for Injection in Subjects With Malignant Plasma Cell Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2934-I-02
Record Dates: First submitted 2025-09-09; First posted 2025-09-18 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Injections, Subcutaneous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2934 injection (subcutaneous injection) (Experimental): Subcutaneous injection，40mg.60mg each time,Cycle 1-3, once a week，Cycle 4-6, once every 2 weeks, if reach PR and above remission after 6 cycles of administration, once every 4 weeks,28 days as a treatment cycle.
  Interventions: Drug: TQB2934 injection (subcutaneous injection)

INTERVENTIONS:
Drug: TQB2934 injection (subcutaneous injection) — TQB2934 is an anti-CD3(Early T Cell Marker)×BCMA (B cell maturation antigen)double-specific antibody，and the isoform is Native Immunoglobulin G1 ( IgG1), which at one end binds to the CD3 receptor on the surface of T cells ,and the other end binds to BCMA(B cell maturation antigen) to recruit T cells around BCMA-positive cells, which can activate T cells .Active T cells release granzyme and perforin to kill BCMA-positive target cells.

SUMMARY:
TQB2934 is an anti-Cluster of Differentiation 3 (CD3) (Early T Cell Marker)×B cell maturation antigen (BCMA) double-specific antibody，and the isoform is IgG1(Native Immunoglobulin G1), which at one end binds to the CD3 receptor on the surface of T cells ,and the other end binds to BCMA(B cell maturation antigen) to recruit T cells around BCMA-positive cells, which can activate T cells .Active T cells release granzyme and perforin to kill BCMA-positive target cells.

TQB2934 for injection (subcutaneous injection) is intended for the treatment of patients with multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily joined the study, signed an informed consent form, and had good compliance;
* 18 years old≤age≤75 years old (calculated based on the date of signing the informed consent); Eastern Cooperative Oncology Group Performance Status (ECOG) score 0~2 points; expected survival is greater than 12 weeks;
* Subjects with multiple myeloma must meet: 1) have a diagnostic record and meet the International Myeloma Working Group Relapsed (IMWG) diagnostic criteria; 2) there is a measurable lesion; 3) Refractory Multiple Myeloma (RRMM) has received at least one line of treatment, and at least one proteasome inhibitor (PI), an immunomodulator (IMiD) and a Cluster of Differentiation 38 (CD38) monoclonal antibody are refractory; 4) disease progression within 12 months after the last treatment or treatment;
* Laboratory inspection standards that meet the program requirements;
* Women of childbearing age should agree that effective contraception must be adopted during the study period and within 6 months after the end of the study, and that serum or urine pregnancy tests will be negative within 7 days before the study enrollment; men should agree that effective contraception must be adopted within 6 months after the end of the study period;

Exclusion Criteria:

* Diagnosed with amyloidosis, active plasma cell leukemia (PCL, peripheral plasma cell proportion ≥5%, or absolute peripheral plasma cell count ≥0.5×109/L), Fahrenheit macroglobulinemia (WM) or POEMS syndrome and other plasma cell tumors;
* Have received allogeneic hematopoietic stem cell transplantation within 1 year before the first medication, or have received autologous hematopoietic stem cell transplantation (ASCT) within 12 weeks before the first medication;
* Those who are known to have invasion of meninges or central nervous system or are highly suspected of invasion of meninges or central nervous system but cannot be identified;
* Have received CD3×BCMA dual anti-anti-treatment in the past;
* Cumulative treatment of dexamethasone >160 mg or equivalent dose of other glucocorticoids within 4 weeks before the first medication, or received targeted therapy, cytotoxic drugs or any antibody therapy within 3 weeks before the first medication, or received proteasome inhibitor therapy or radiotherapy within 2 weeks before the first medication, or received immunomodulatory therapy within 1 week before the first medication;
* Those who have received Chinese patent medicine treatments within 2 weeks before the first medication have received National Medical Products Administration (NMPA) -approved drug instructions that clearly have anti-tumor indications;
* Those who have a history of live attenuated vaccination within 4 weeks before the first medication or plan to undergo live attenuated vaccination during the study period;
* A person with a history of severe allergies of unknown causes, or known to be allergic to monoclonal antibody drugs or exogenous human immunoglobulin, or known to be allergic to TQB2934 for injection or excipients in drug preparations;
* Have appeared within 3 years before the first medication or are currently suffering from other malignant tumors;
* Unrelieved toxic reactions above Common Terminology Criteria (CTC) AE level 1 caused by any previous treatment, excluding hair loss, fatigue and peripheral neuropathy;
* Those who have received major surgical treatment, obvious traumatic injury or expected research treatment within 4 weeks before the first medication, or have long-term uncured wounds or fractures;
* Arterial/venous thrombosis events occurred within 6 months before the first dose;
* People with a history of abuse of psychotropic substances and cannot quit or have mental disorders, or suffer from epilepsy and need treatment;
* Those with poor blood pressure control;
* People with poor diabetes control;
* People with severe bacterial, viral or systemic fungal infections that are active or uncontrollable within 4 weeks before the first medication;
* People with hepatitis or decompensated cirrhosis;
* People with active tuberculosis, a history of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonia, radioactive pneumonia that needs treatment, or active pneumonia with clinical symptoms;
* People who have had or are currently suffering from asthma within 2 years before the first medication, or who have chronic obstructive pulmonary disease (COPD) and have a forceful exhalation volume (FEV1) in the first second <50% expected value;
* Those who have had asthma within 2 years before the first medication or are currently suffering from asthma;
* People suffering from major cardiovascular diseases;
* Have a history of immunodeficiency;
* According to the researcher's judgment, there are concomitant diseases that seriously endanger the safety of the subject or affect the completion of the study, or subjects who believe there are other reasons that are not suitable for enrollment;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Peak time (Tmax) | Within 120 hours after administration
  It refers to the time when TQB2934 (subcutaneous injection) is administered for injection to reach the maximum blood drug concentration.
Peak drug concentration (Cmax) | Within 120 hours after administration
  It refers to the highest blood drug concentration after administration of TQB2934 (subcutaneous injection).
Area under the plasma concentration-time curve (AUC0-last) | Within 120 hours after administration
  To characterize the pharmacokinetics of TQB2934 by assessment of area under the plasma concentration time curve.
Elimination half-life (t1/2) | Within 120 hours after administration
  t1/2 is time it takes for the blood concentration of TQB2934 to drop by half.
Apparent clearance (CL) | Within 120 hours after administration
  Apparent clearance (CL)
Adverse events(AEs) | Up to 24 months
  Incidence and severity of subjects with adverse events(AEs), Abnormal laboratory test value and serious adverse events

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 24 months
  Proportion of subjects with best response as Partial relief (PR), Very good partial relief (VGPR), Complete Response (CR), Strict Complete Response (sCR)
Clinical benefit rate (CBR) | Up to 24 months
  Proportion of subjects with best response as Minor relief (MR), PR(Partial relief), VGPR(Very good partial relief), CR (Complete Response), sCR (Strict Complete Response)
very good partial response rate (VGPR) | Up to 24 months
  Proportion of subjects whose best response is VGPR, CR, sCR;
Complete Response (CR) Rate | Up to 24 months
  Proportion of subjects whose best response is CR
Strict Complete Response (sCR) | Up to 24 months
  Proportion of subjects whose best response is sCR;
Negative rate of minimal residual disease (MRD) | Up to 24 months
  The proportion of subjects with negative MRD (<10-5, multicolor flow cytometry or next-generation sequencing) at any time point from the first administration of the trial drug to disease progression or before receiving new anti-tumor therapy;
Duration of remission (DOR) | Up to 24 months
  For all subjects whose best response was PR, VGPR, CR, sCR, the time from the date of first achieving PR, VGPR, CR, sCR to the date of first definite disease progression or (any cause) death(whichever occurs first).
Time to first remission (TTR) | Up to 24 months
  Among all the subjects whose best response is PR, VGPR, CR, sCR, the time from the first administration of the test drug to the date of the first PR and above remission.
Progression-free survival (PFS) | Up to 24 months
  The time between the first dose of the trial drug and the date of first definite disease progression or death (from any cause), whichever occurs first.
Overall survival (OS) | Up to 24 months
  Time from first dose of study drug to date of death from any cause.
Antidrug antibody (ADA) incidence and changes over time | Up to 24 months
  Positive incidence of anti-drug antibodies and changes over time

CONTACTS AND LOCATIONS:
Locations (14):
- China (14):
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The Affiliated Hospital of Chengde Medical College, Chengde, Hebei
  - North China University of Science and Technology Affiliated Hospital, Tangshan, Hebei
  - Nanjing Drum Tower hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Nanchang University First Affiliated Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Heze Municipal Hospital, Heze, Shandong
  - Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality